CLINICAL TRIAL: NCT05912855
Title: To Investigate the Impact of Analgesic Management Guided by qNOX Monitoring on the Comfort and Prognosis of Mechanically Ventilated ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Other Study IDs: GWang009
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPS（Behavioral Pain Scale）and physiological index monitoring guided analgesia group
- Analgesia group guided by qNOX
  Interventions: Device: qNOX

INTERVENTIONS:
Device: qNOX — Non
  Groups: Analgesia group guided by qNOX

SUMMARY:
Purpose: To explore the effect of analgesic management under the guidance of qNOX monitoring on the comfort level and prognosis of patients with mechanical ventilation in ICU.

Method:After admission to ICU, the patients were randomly divided into the analgesia group guided by BPS（Behavioral Pain Scale） and physiological indicators monitoring and qNOX-guided analgesia group (qNOX group). Sedation and analgesia program after admission to ICU (continuous injection pump) : propofol 1.5-4.5mg/kg.h, remifentanil 5-8ug/kg.h, maintain sedation goals RASS（Richmond Agitation-Sedation Scale）-3 to -4 scores, BPS（Behavioral Pain Scale）3 to 4 scores. The researchers worked with the bedside nurse to plan different care procedures, including :1) central venous catheter or arterial catheter puncture; 2) The patient is turned over completely so that the back can be washed and the sheets changed; 3) Endotracheal sputum aspiration (patients with intubation or in tracheotomy state ); 4) Dressing the wound.

Primary outcome:Value of qNOX at BPS（Behavioral Pain Scale）≥5 (qNOX sensitivity, specificity, positive predictive value and negative predictive value) Secondary outcome:To investigate the patient baseline variables that may affect qNOX; Variables that may influence qNOX in relation to critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older who are undergoing abdominal, orthopedic, ENT（ear-nose-throat）, urological, neurosurgical or cardiothoracic surgery and require ICU treatment with mechanical ventilation while having an RASS（Richmond Agitation-Sedation Scale）-3 or -4 score;
2. Patients unable to self-assess pain intensity using NRS（Numerical Pain Rating Scale）;
3. Patients who have provided informed consent.

Exclusion Criteria:

1. < 18 years of age;
2. Pregnant individuals;
3. Patients with communication impairments, such as those who have experienced cerebrovascular accidents;
4. A decision to withdraw life-sustaining treatment or an unstable medical condition that disrupts planned routine care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients receiving mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Value of qNOX with BPS≥5 | During procedure
  Sensitivity, specificity, positive predictive value and negative predictive value of qNOX.